CLINICAL TRIAL: NCT02531568
Title: A Phase I, Open-label, Single-Centre, Drug-Drug Interaction Study to Evaluate the Influence of MT-3995 on Pharmacokinetics(PK) and Pharmacodynamics of Warfarin in Healthy Subjects
Brief Title: Drug Interaction Study of Warfarin and MT-3995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: MT-3995-E10
Record Dates: First submitted 2015-08-04; First posted 2015-08-24 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — Warfarin; apararenone

ARMS (1):
- Warfarin and MT-3995 (Experimental): Subjects will be administered a single dose of warfarin on day1. Subjects will be administered MT-3995 Days 8 to 20. Subjects will be administered MT-3995 and warfarin on Day21. Subjects will be administered MT-3995 from Day 22 to 27.
  Interventions: Drug: Warfarin; Drug: MT-3995

INTERVENTIONS:
Drug: Warfarin
Drug: MT-3995

SUMMARY:
The purpose of this study is to evaluate the effects of MT-3995 on the PK of warfarin

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the potential effects of multiple once daily doses of MT-3995 on the PK of (S)-warfarin and (R)-warfarin after single-dose administration of racemic warfarin

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent to participate in this study
* Healthy, free from clinically significant illness or disease
* White Caucasian male or female, aged 18 to 55 years
* Body weight ranging from 50 (females) and 60 (males) to110 kg (inclusive)
* Must have coagulation test results (including international normalised ratio [INR] and activated partial thromboplastin time [aPTT]) within the laboratory reference range at Screening.

Exclusion Criteria:

* Presence or history of serious adverse reaction or allergy to any medicinal product
* Known contraindication or adverse reaction to warfarin.
* Presence of Cytochrome P450 2C9 (CYP2C9) and Vitamin K epoxide reductase complex subunit 1 (VKORC1) genetic polymorphisms that are known to increase warfarin sensitivity at Screening.
* Known contraindications to heparin administration.
* Known contraindication to parenteral vitamin K administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cmax of warfarin with MT-3995 versus warfarin alone | 8 days
AUC of warfarin with MT-3995 versus warfarin alone | 8 days

SECONDARY OUTCOMES:
International normalized ratio (INR) max of warfarin with MT-3995 versus warfarin alone | 8 days
INR AUC of warfarin with MT-3995 versus warfarin alone | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Horst Heuer, Dr, Principal Investigator — Nuvisan GmbH
Locations (1):
- Clinical research organization, Neu-Ulm, Wegenerstraße, Germany

REFERENCES:
- [Derived] Nakamura T, Shimizu H, Kawaguchi A. Drug-Drug Interactions of the Nonsteroidal Mineralocorticoid Receptor Antagonist Apararenone With Midazolam, Warfarin, and Digoxin: A Phase 1 Studies in Healthy Volunteers. Clin Ther. 2020 Nov;42(11):2171-2183.e4. doi: 10.1016/j.clinthera.2020.09.002. Epub 2020 Nov 3. PMID 33153727